CLINICAL TRIAL: NCT01674166
Title: A Single-dose Pharmacokinetic Trial of 0.03 mg/kg R108512 Solution in Paediatric Subjects, Aged >= 4 to <= 12 Years With Functional Faecal Retention (FFR).
Brief Title: Single Dose Pharmacokinetics of Prucalopride in Paediatric Subjects, With Functional Faecal Retention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRU-USA-12
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-06

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — prucalopride

ARMS (1):
- prucalopride (Experimental): single dose 0.03 mg/kg prucalopride open label
  Interventions: Drug: prucalopride

INTERVENTIONS:
Drug: prucalopride — single dose 0.03 mg/kg prucalopride open label

SUMMARY:
The purpose of this study is characterize the pharmacokinetics of a single oral dose of 0.03 mg/kg prucalopride in paediatric subjects aged >= 4 to <= 12 years with functional faecal retention.

Hypothesis:

Pharmacokinetic profile of prucalopride in paediatric subjects is expected to resemble the adult pharmacokinetic profile

DETAILED DESCRIPTION:
This is a multicentre, open-label, single-dose pharmacokinetic trial. A minimum of 24 paediatric subjects (aged ≥ 4 to ≤ 12 years) with functional faecal retention (FFR) were administered a single dose of prucalopride in oral solution.

All subjects who qualified to enter the trial received a single dose of 0.03 mg/kg prucalopride oral solution at Hour 0 on Day 1. One blood sample was drawn prior to dosing, and 13 samples were drawn over the 72-hour interval following the single dose or prucalopride. Urine was collected quantitatively for the first 24 hours. Plasma prepared from blood samples and urine samples were assayed for prucalopride concentrations. Safety was monitored over the 72-hour interval following the dose of trial medication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed diagnosis of FFR, defined as a minimum 2-month history of faecal impaction, plus at least one of the following:

  * < 3 bowel movements per week at the toilet;
  * A history of soiling;
* Male and female subjects ≥ 4 to ≤ 12 years of age, with a Tanner stage 1 of 2 or less;
* Weight-height proportionality for age within the 5th and 95th percentile;
* Written informed consent, signed by the subject's legal guardian and by the investigator, and;
* Subject assent documented in the form of a note-to-file in the subject's source documentation.

Exclusion Criteria:

* Requirement for any medication during the period of the trial;
* Evidence by examination or laboratory tests of abnormal growth;
* An abnormal neurologic examination;
* Cystic fibrosis;
* History of, or current anorectal malformations;
* Diagnosed chromosomal abnormalities (e.g., Down's Syndrome);
* Disease state or surgery known to significantly affect the gastrointestinal absorption of drugs, or the assessment of the trial drug's effect;
* Any history, clinical and/or biochemical evidence of clinically significant renal or liver disease or cirrhosis;
* Clinically significant anaemia;
* Use of any investigational drug within the 4-week period prior to administration of trial medication.

Ages: 4 Years to 12 Years
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 1998-11; Primary Completion 1999-05 (Actual); Study Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of a single oral dose of 0.03 mg/kg prucalopride in paediatric subjects aged >= 4 to <= 12 years with functional faecal retention.

SECONDARY OUTCOMES:
Secondary efficacy variables: safety and tolerability of a single dose of prucalopride 0.03 mg/kg given to paediatric subjects with FFR.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Winter, M.D., Principal Investigator — Massachusetts General Hospital for Children, Boston, Massachusetts, USA

REFERENCES:
- [Derived] Winter HS, Di Lorenzo C, Benninga MA, Gilger MA, Kearns GL, Hyman PE, Vandeplassche L, Ausma J, Hoppenbrouwers M. Oral prucalopride in children with functional constipation. J Pediatr Gastroenterol Nutr. 2013 Aug;57(2):197-203. doi: 10.1097/MPG.0b013e318292f9ea. PMID 23535761